CLINICAL TRIAL: NCT02263001
Title: Auricular Acupuncture Therapy for Treatment of Musculoskeletal Pain in the Setting of Military Personnel: A Randomized Trial
Brief Title: Acupuncture Therapy for Treatment of Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Scripps Center for Integrative Medicine (Other); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul J. Mills, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMCSD.2011.0119
Record Dates: First submitted 2014-10-03; First posted 2014-10-13 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Musculoskeletal Pain
Keywords: Auricular therapy; Acupuncture; Acute, sub-acute pain; Auricular Acupuncture Needles
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Auricular Acupuncture Plus Usual Care (Experimental): Auricular acupuncture therapy for treatment of musculoskeletal pain, plus usual care therapy consisting of over-the-counter and prescribed pharmacotherapy.
  Interventions: Other: Auricular acupuncture
- Usual Care Only (Active Comparator): Usual care therapy for treatment of musculoskeletal pain. Usual care therapy consists of over-the-counter and prescribed pharmacotherapy.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Auricular acupuncture — Auricular therapy for treatment of musculoskeletal pain
  Arms: Auricular Acupuncture Plus Usual Care
Other: Usual Care — Usual care therapy consists of over-the-counter and prescribed pharmacotherapy
  Arms: Usual Care Only

SUMMARY:
Musculoskeletal injuries resulting in pain are one of the most common reasons for disability and missed duty among military personnel. Additionally, these injuries may create impairment in the area of optimal function, sleep and mood that may not be completely resolved with currently available therapies. This scenario creates the setting for testing and incorporation of additional treatment options to potentially improve care outcomes. Recent investigations have examined the adjunctive use of auricular therapy, which utilizes various interventions, typically needle-based, to stimulate the ear. This intervention appears to modulate the autonomic nervous system to produce more rapid onset of pain relief and reduction in pain related co-morbidities. For this trial of adjunctive auricular therapy, active duty personnel presenting with an acute or sub-acute musculoskeletal injury triaged to outpatient care for treatment will be studied. Subjects randomized to auricular treatment will receive, in addition to standard care, up to 12 treatments over a maximum of 3 months from a clinician trained in auricular therapy. This trial will specifically examine whether the addition of a specific auricular therapy protocol to standard care will have a beneficial impact on the pain and functionality of military personnel who sustain an acute or sub-acute musculoskeletal injury.

DETAILED DESCRIPTION:
Musculoskeletal injuries resulting in pain are one of the most common reasons for disability and missed duty among military personnel. Additionally, these injuries may create impairment in the area of optimal function, sleep and mood that may not be completely resolved with currently available therapies. This scenario creates the setting for testing and incorporation of additional treatment options to potentially improve care outcomes. Recent investigations have examined the adjunctive use of auricular therapy, which utilizes various interventions, typically needle-based, to stimulate the ear. This intervention appears to modulate the autonomic nervous system to produce more rapid onset of pain relief and reduction in pain related co-morbidities. For this trial of adjunctive auricular therapy, 150 subjects will be enrolled at the Naval Medical Center San Diego. Subjects will be active duty personnel aged 18-60 years old presenting with an acute or sub-acute musculoskeletal injury triaged to outpatient care for treatment. Subjects randomized to auricular treatment will receive, in addition to standard care, up to 12 treatments over a maximum of 3 months from a clinician trained in auricular therapy. This trial will specifically examine whether the addition of a specific auricular therapy protocol to standard care will have a beneficial impact on the pain and functionality of military personnel who sustain an acute or sub-acute musculoskeletal injury.

ELIGIBILITY:
Inclusion Criteria:

* Active duty personnel with a musculoskeletal injury
* Injuries eligible for inclusion include all acute or subacute (<3 months in duration) non-fracture related musculoskeletal injuries of the axial or peripheral skeleton
* Examples of injuries meeting inclusion include acute or sub-acute injuries of the neck, low back as well as the upper and lower extremities
* Individuals with the pre-existing chronic pain pain greater than 3 months in duration will be eligible if they have a presenting acute or sub-acute pain condition as described above

Exclusion Criteria:

* Injuries involving hospitalization or surgery for treatment in the presenting area of pain
* Rheumatologic and autoimmune conditions which may be creating pain, such as rheumatoid arthritis, advanced osteoarthritis, or spinal stenosis
* Contra-indication to needle use including known bleeding disorder and psychogenic issues related to needle use (needle-phobia)"
* Evidence or history of clinically significant immune deficiency, hematological, oncological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or severe allergic disease (including to metals and adhesive tapes) which could interfere with this study
* Individuals with progressive radiating pain with motor-sensory changes (including weakness or numbness) related to their presenting pain complaint
* Any contra-indication to the use of electrical stimulation, including history of epilepsy, cardiac arrhythmias, pacemaker or any other implantable programmable device
* Treatment with acupuncture or auricular therapy within the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary musculoskeletal pain | 12 weeks
  Standardized scales and clinical assessments to determine if the addition of AT will significantly decrease pain at noted time endpoints after initiation of treatment compared to UC.

SECONDARY OUTCOMES:
Musculoskeletal pain related to co-morbities | 12 weeks
  Standardized scales and clinical assessments to determine if the addition of AT will significantly improve pain related co-morbidities (based on the 0-10 BPI Pain interference scale and SF-8) at noted endpoints after initiation of treatment than UC.
Return of functional ability | 12 weeks
  Standardized scales and clinical assessments to determine if the addition of AT will significantly improve functionality at noted endpoints after initiation of treatment vs. UC.
Reduction of pain medication use | 12 weeks
  Assessment of pharmacy records and self report to determine if AT will provide significant reduction in need for pain medication as compared to UC.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bonakdar, MD, Principal Investigator — Scripps Integrative Medical Center, La Jolla, CA
Locations (1):
- Naval Medical Center San DIego, San Diego, California, United States